CLINICAL TRIAL: NCT05331768
Title: Comparison of Endoscopic Band Ligation Plus 24-hour Versus 72-hour Terlipressin Therapy for the Control of Acute Variceal Bleeding in Patients With Liver Cirrhosis at a Tertiary Center in Mexico
Brief Title: Comparison of Endoscopic Band Ligation Plus 24-hour Versus 72-hour Terlipressin Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Clinical Professor, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Terlipressin proyect
Record Dates: First submitted 2022-03-29; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Esophageal and Gastric Varices
Keywords: Terlipressin; Liver Cirrhosis; Esophageal and Gastric Varices,; Collateral Circulations
MeSH Terms: conditions — Esophageal and Gastric Varices; Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: This was a randomized clinical trial. Eligible patients were randomised to receive banding ligation plus terlipressin infusion for 24 hours or banding ligation plus terlipressin infusion for 72 hours
Who Masked: Participant
Masking Description: Subjects were randomly allocated to banding ligation plus terlipressin infusion for 24 hours (24-h group) or banding ligation plus terlipressin infusion for 72 hours (72-h group) using a blocked allocation strategy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 24-h group (Experimental): The 24-h group received intravenous terlipressin (Glypressin® Ferring Pharmaceuticals) as an initial intravenous bolus of 2 mg (10 ml) and thereafter every 6 hours for a period of 24 hours.
  Interventions: Combination Product: banding ligation plus terlipressin infusion
- 72-h group (Active Comparator): The 72-h group received the standard treatment with administration of intravenous terlipressin (Glypressin® Ferring Pharmaceuticals) with an initial intravenous bolus of 2 mg (10 ml) and thereafter every 6 hours for a period of 72 hours. Terlipressin was administered blinded after endoscopic treatment and infused as a 5 ml bolus in a pre-prepared syringe
  Interventions: Combination Product: banding ligation plus terlipressin infusion

INTERVENTIONS:
Combination Product: banding ligation plus terlipressin infusion — Subjects were randomly allocated to banding ligation plus terlipressin infusion for 24 hours (24-h group) or banding ligation plus terlipressin infusion for 72 hours (72-h group) using a blocked allocation strategy. The 72-h group received the standard treatment with administration of intravenous terlipressin (Glypressin® Ferring Pharmaceuticals) with an initial intravenous bolus of 2 mg (10 ml) and thereafter every 6 hours for a period of 72 hours. Terlipressin was administered blinded after endoscopic treatment and infused as a 5 ml bolus in a pre-prepared syringe. The 24-h group received intravenous terlipressin (Glypressin® Ferring Pharmaceuticals) as an initial intravenous bolus of 2 mg (10 ml) and thereafter every 6 hours for a period of 24 hours.

SUMMARY:
In the Western world, liver cirrhosis is a significant issue. Acute variceal bleeding (AVB) is a considerable complication of cirrhosis associated with high mortality. Still, the combination of endoscopic variceal ligation and terlipressin-like treatment decreases the risks of rebleeding and mortality. This therapy with terlipressin usually was used for 72 hours. However, there are some studies demostrating that using terlipressin for 24 hours could control variceal bleeding with fewer side effects.

DETAILED DESCRIPTION:
In the Western world, liver cirrhosis is a significant issue. Acute variceal bleeding (AVB) is a considerable complication of cirrhosis associated with high mortality. Still, the combination of endoscopic variceal ligation and terlipressin-like treatment decreases the risks of rebleeding and mortality. This therapy with terlipressin usually was used for 72 hours. However, there are some studies demostrating that using terlipressin for 24 hours could control variceal bleeding with fewer side effects.

Objective: To compare endoscopic band ligation plus terlipressin for 24 vs 72 hours during acute variceal bleeding in liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years and older
* Both genders,
* Diagnosis of liver cirrhosis with a Child-Pugh score ≤ 11 (class B or C)
* Acute variceal bleeding were included

Exclusion Criteria:

* Patients with contraindications to terlipressin (pregnancy, breastfeeding, or severe cardiopulmonary diseases),
* Presence of sepsis,
* Multi-organ failure,
* The requirement of continuous ionotropic or ventilatory support,
* Bleeding disorders,
* Hepatocellular carcinoma or other extrahepatic malignanc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Compare the 24-h group vs 72-h group | The total study time ranges from the first day of telmipressin infusion to 6 weeks after the event
  Differences between groups at baseline were evaluated with Student's t-test test for continuous variables and proportions were compared using the Chi2 or Fisher test.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro González-Ojeda, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Centro Médico Nacional de Occidente, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
It is expected to find a journal that is interested in our research and that is open access

REFERENCES:
- [Background] Roesch-Dietlen F, Gonzalez-Santes M, Sanchez-Maza YJ, Diaz-Roesch F, Cano-Contreras AD, Amieva-Balmori M, Garcia-Zermeno KR, Salgado-Vergara L, Remes-Troche JM, Ortigoza-Gutierrez S. Influence of socioeconomic and cultural factors in the etiology of cirrhosis of the liver. Rev Gastroenterol Mex (Engl Ed). 2021 Jan-Mar;86(1):28-35. doi: 10.1016/j.rgmx.2020.01.002. Epub 2020 Apr 25. English, Spanish. PMID 32345507
- [Background] Berardo C, Di Pasqua LG, Cagna M, Richelmi P, Vairetti M, Ferrigno A. Nonalcoholic Fatty Liver Disease and Non-Alcoholic Steatohepatitis: Current Issues and Future Perspectives in Preclinical and Clinical Research. Int J Mol Sci. 2020 Dec 17;21(24):9646. doi: 10.3390/ijms21249646. PMID 33348908
- [Background] Boregowda U, Umapathy C, Halim N, Desai M, Nanjappa A, Arekapudi S, Theethira T, Wong H, Roytman M, Saligram S. Update on the management of gastrointestinal varices. World J Gastrointest Pharmacol Ther. 2019 Jan 21;10(1):1-21. doi: 10.4292/wjgpt.v10.i1.1. PMID 30697445
- [Background] Bosch J, Pizcueta MP, Fernandez M, Feu F, Cirera I, Luca A, Garcia-Pagan JC. Hepatic, splanchnic and systemic haemodynamic abnormalities in portal hypertension. Baillieres Clin Gastroenterol. 1992 Sep;6(3):425-36. doi: 10.1016/0950-3528(92)90030-i. PMID 1421593
- [Background] Kalambokis G, Tsiouris S, Tsianos EV, Baltayiannis G, Pakou B, Fotopoulos A. Effects of terlipressin and somatostatin on liver and thorax blood volumes in patients with cirrhosis. Liver Int. 2010 Oct;30(9):1371-8. doi: 10.1111/j.1478-3231.2010.02322.x. PMID 20738780
- [Background] Kovalak M, Lake J, Mattek N, Eisen G, Lieberman D, Zaman A. Endoscopic screening for varices in cirrhotic patients: data from a national endoscopic database. Gastrointest Endosc. 2007 Jan;65(1):82-8. doi: 10.1016/j.gie.2006.08.023. PMID 17185084
- [Background] Garcia-Tsao G, Sanyal AJ, Grace ND, Carey W; Practice Guidelines Committee of the American Association for the Study of Liver Diseases; Practice Parameters Committee of the American College of Gastroenterology. Prevention and management of gastroesophageal varices and variceal hemorrhage in cirrhosis. Hepatology. 2007 Sep;46(3):922-38. doi: 10.1002/hep.21907. No abstract available. PMID 17879356
- [Background] Fortune BE, Groszmann RJ. Combination of splanchnic vasoconstrictors and endoscopic band ligation is an effective treatment strategy for acute variceal hemorrhage; but how do we get those drugs approved by the FDA? Hepatology. 2014 Sep;60(3):789-91. doi: 10.1002/hep.27080. Epub 2014 Jul 28. No abstract available. PMID 24700393
- [Background] Bendtsen F, Krag A, Moller S. Treatment of acute variceal bleeding. Dig Liver Dis. 2008 May;40(5):328-36. doi: 10.1016/j.dld.2007.12.005. Epub 2008 Feb 1. PMID 18243077
- [Background] Zhou X, Tripathi D, Song T, Shao L, Han B, Zhu J, Han D, Liu F, Qi X. Terlipressin for the treatment of acute variceal bleeding: A systematic review and meta-analysis of randomized controlled trials. Medicine (Baltimore). 2018 Nov;97(48):e13437. doi: 10.1097/MD.0000000000013437. PMID 30508958
- [Background] Banares R, Albillos A, Rincon D, Alonso S, Gonzalez M, Ruiz-del-Arbol L, Salcedo M, Molinero LM. Endoscopic treatment versus endoscopic plus pharmacologic treatment for acute variceal bleeding: a meta-analysis. Hepatology. 2002 Mar;35(3):609-15. doi: 10.1053/jhep.2002.31354. PMID 11870374
- [Background] Krag A, Borup T, Moller S, Bendtsen F. Efficacy and safety of terlipressin in cirrhotic patients with variceal bleeding or hepatorenal syndrome. Adv Ther. 2008 Nov;25(11):1105-40. doi: 10.1007/s12325-008-0118-7. PMID 19018483
- [Background] Dohler KD, Walker S, Mentz P, Forssmann K, Staritz M. [Vasoconstrictive Therapies for Bleeding Esophageal Varices and their Mechanisms of Action]. Z Gastroenterol. 2003 Oct;41(10):1001-16. doi: 10.1055/s-2003-42931. German. PMID 14562199
- [Background] Salim A, Malik K, Haq IU, Butt AK, Alam A. Comparison of 12-Hour with 72-Hour Terlipressin Therapy for Bleeding Esophageal Varices. J Coll Physicians Surg Pak. 2017 Jun;27(6):334-337. PMID 28689520
- [Background] Moller S, Hansen EF, Becker U, Brinch K, Henriksen JH, Bendtsen F. Central and systemic haemodynamic effects of terlipressin in portal hypertensive patients. Liver. 2000 Feb;20(1):51-9. doi: 10.1034/j.1600-0676.2000.020001051.x. PMID 10726961
- [Background] Yao Q, Chen W, Yan C, Yu J, Jiang T, Cao H. Efficacy and Safety of Treatments for Patients With Portal Hypertension and Cirrhosis: A Systematic Review and Bayesian Network Meta-Analysis. Front Med (Lausanne). 2021 Sep 3;8:712918. doi: 10.3389/fmed.2021.712918. eCollection 2021. PMID 34540867
- [Background] Abid S, Jafri W, Hamid S, Salih M, Azam Z, Mumtaz K, Shah HA, Abbas Z. Terlipressin vs. octreotide in bleeding esophageal varices as an adjuvant therapy with endoscopic band ligation: a randomized double-blind placebo-controlled trial. Am J Gastroenterol. 2009 Mar;104(3):617-23. doi: 10.1038/ajg.2008.147. Epub 2009 Feb 17. PMID 19223890
- [Background] Ioannou G, Doust J, Rockey DC. Terlipressin for acute esophageal variceal hemorrhage. Cochrane Database Syst Rev. 2003;(1):CD002147. doi: 10.1002/14651858.CD002147. PMID 12535432
- [Background] Yeh JH, Lo GH, Huang RY, Lin CW, Wang WL, Perng DS. Short-course vasoconstrictors are adequate for esophageal variceal bleeding after endoscopic variceal ligation: A systematic review and meta-analysis. Sci Prog. 2021 Jul-Sep;104(3):368504211031711. doi: 10.1177/00368504211031711. PMID 34260315
- [Background] Azam Z, Hamid S, Jafri W, Salih M, Abbas Z, Abid S, Shah H. Short course adjuvant terlipressin in acute variceal bleeding: a randomized double blind dummy controlled trial. J Hepatol. 2012 Apr;56(4):819-24. doi: 10.1016/j.jhep.2011.11.019. Epub 2011 Dec 16. PMID 22178268
- [Result] Byrne CD, Targher G. NAFLD: a multisystem disease. J Hepatol. 2015 Apr;62(1 Suppl):S47-64. doi: 10.1016/j.jhep.2014.12.012. PMID 25920090